CLINICAL TRIAL: NCT01294488
Title: Using Technology to Augment the Implementation and Effectiveness of PCIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-5085
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Child Externalizing Problems
Keywords: PCIT; Child Maltreatment Prevention; Practitioner Fidelity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phone Consultation (Experimental): Therapists receive phone consultation for 6 months during the course of the project.
  Interventions: Behavioral: Parent-Child Interaction Therapy
- Remote Real-Time Consultation (Experimental): Therapists receive consultation for 6 months via polycommunication technology.
  Interventions: Behavioral: Parent-Child Interaction Therapy

INTERVENTIONS:
Behavioral: Parent-Child Interaction Therapy — Therapists receive training in Parent-Child Interaction Therapy (PCIT) and receive supervision in their implementation of PCIT skills via phone consultation and polycommunication technology, each for 6 months.

SUMMARY:
The overarching aim of the proposed study is to test the implementation effectiveness of two implementation approaches-Remote Real-Time (RRT) using the internet telemedicine technology and traditional Phone Consultation (PC) for training practitioners in PCIT. The study will add to emerging knowledge about how technology can facilitate the transport of evidence-based intervention models into field settings.

DETAILED DESCRIPTION:
Parent-Child Interaction Therapy (PCIT) is an empirically supported behavioral parent training program for reducing aggressive behavior in young children and for reducing future rates of child physical abuse. Prior research has found that an adapted version of PCIT developed specifically for violent parents in the child welfare system reduced future child physical abuse recurrence rates from 49% to 19%. OUHSC/CCAN researchers, in prior and ongoing studies, have found the benefits of PCIT to be durable over time and to generalize across settings and across children in the same family. Culturally-specific adaptations of PCIT and adaptations for older abused children and their abusive parents have been developed. A number of blue-ribbon panels have recommended PCIT for widespread dissemination in child abuse prevention and intervention service systems, but uptake of PCIT has been limited. One reason for this is that the traditional PCIT practitioner training models are not easily replicable in field settings. PCIT has historically been taught in University-based training programs (graduate programs, internships, etc.) and includes several months of co-therapy mentoring where trainers work directly with trainees during live sessions. In contrast, given the difficulties of conducting co-therapy mentoring in field settings, training for widespread implementation has generally involved initial training in the model followed by phone consultation.

OUHSC/CCAN researchers have pilot- and feasibility tested a system using internet-based telemedicine technology to deliver live, mentored PCIT training. OUHSC/CCAN researchers have piloted Remote Real-Time (RRT) training at sites in Utah, Seattle, Alaska, Oregon, and Oklahoma. Feasibility appears excellent, and the approach has been well received. Moreover, RRT implementation revealed misapplications of the model that had gone unaddressed in phone consultation. This research project will make use of planned, funded PCIT start-up implementations at 20-24 agency sites in Washington and Oklahoma. Study participants will include agency practitioners engaged in implementing the PCIT model and families receiving PCIT services at these community agencies. Using a multilevel interrupted time series randomized design; the study will compare the RRT implementation approach with standard phone consultation (PC). Outcomes will include practitioner fidelity and competency in implementing PCIT, practitioner acceptance and satisfaction with PCIT, and family outcomes of parental skill acquisition, parent satisfaction, child aggressive and oppositional behaviors, and rates of future child welfare abuse reports. A mediational model is proposed in which differences in client outcomes are mediated by improved practitioner fidelity and competency. Cost effectiveness and practitioner response to the implementation approach will be examined. The study thus will inform strategies for facilitating widespread dissemination and implementation with fidelity of the evidence-based PCIT model, thereby making the model available to a broader range of agencies and practitioners working with at-risk families.

ELIGIBILITY:
Inclusion Criteria:

A major inclusion criterion for agencies is existing plans and financial support for PCIT implementation because this study's resources cannot fund the phase one didactic training or clinical implementation. The proposed agencies all have existing funding, including demonstration grants, Children's Justice grant funding, state contracts, federal implementation funding, Indian Health Services funding, or SAMHSA funding specifically to support their PCIT implementation. However without the current project, none of the agency sites proposed for this study would be using RRT or assessing therapist fidelity; this study thus provides quality assurance mechanisms that would be unavailable otherwise. The agencies have reviewed and agreed to a set of agency inclusion criteria for study participation:

* The agency should be committed to developing a PCIT program, not simply training staff. There should be a commitment by leadership to the program's long-term sustainability, including sustaining the program through staff turn-over.
* The agency should identify a minimum of three staff for PCIT training (with two staff members acceptable from very small agencies that do not have three child service providers), at least one of which is a supervisor. Licensed mental health practitioner staff with a Master's degree or higher are strongly preferred, although exceptions may be made in cases where agencies do not have Master's level staff. (For example, some agencies conducting culturally relevant programs for minority or rural populations are not always able to employ licensed mental health provider staff. Because RRT may be especially salient for some of these agencies, these agencies will not be excluded from the study.)
* The agency should be committed to providing the resources and staff availability to complete the basic PCIT training package, standard PC consultation, and staff participation in approximately six months of RRT training.
* The agency should have or be in the process of developing the physical infrastructure to deliver PCIT. Physical infrastructure includes PCIT rooms with sound equipment, bug-in-the-ear equipment, and video recording equipment.
* The agency will need to have a dedicated broadband internet line for the RRT equipment.
* The agency should be able to demonstrate that it has or will develop a referral network sufficient to provide enough PCIT cases so that therapists can develop mastery. This can include referral commitments and support from local child welfare offices, courts, schools, and so forth. If the agency plans to serve child welfare parents whose children are in foster care, it is imperative that there are firm commitments for a transportation plan. Preliminary work may be necessary to gain the cooperation of child welfare and courts to insure that service plans and court orders are consistent with PCIT (i.e. allowing joint parent-child sessions).
* The agency agrees that basic PCIT training will meet OUHSC training guidelines (to be described later).
* If clients consent to participate, the agency agrees to archive video recordings of all PCIT sessions and basic PCIT clinical measures from clients.
* The agency is in a state that agrees to provide OUHSC with child welfare outcome data.
* In the event the agency's PCIT start-up plan requires that they begin PCIT services prior to the start of the study, they will commence archiving session and client data so that early session fidelity and competency and client outcomes can be tracked. Standard PC consultation will be provided until the study begins. Session- and client-level data are routinely collected as part of PCIT implementation, to guide clinical intervention and assure quality of services. However, no data will be used for research purposes unless therapists and clients provide informed consent for its use.
* The study will retain the right to involuntarily remove an agency and its therapists from the study if PCIT implementation and data collection at the agency proves infeasible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2007-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Child Maltreatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Funderburk, Ph.D., Principal Investigator — OUHSC
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States